CLINICAL TRIAL: NCT00480662
Title: A 6-Month, Multicenter, Double-Blind, Randomized, Active-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Alendronate 280-mg Oral Buffered Solution Once Weekly in Patients With Paget's Disease of Bone
Brief Title: A Research Study to Test the Effectiveness of MK0217 in Patients With Paget's Bone Disease (0217-206)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-206; MK0217-206; 2007_555
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Paget's Disease of Bone
Keywords: Paget's bone disease
MeSH Terms: conditions — Osteitis Deformans | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: alendronate — Duration of Treatment : 6 Months
  Other Names: MK0217

SUMMARY:
To test the safety, effectiveness of MK0217 when taken once a week for six months in treating patients with Paget's bone disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 to 90 years with a diagnosis of Paget's bone disease

Exclusion Criteria:

* Patient cannot stand or sit upright for at least 30 minutes
* Patient has difficulty swallowing or problems with digestive system

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-10; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Patients will have a decrease of at least 30% in their blood alkaline phosphatase level after 6 months

SECONDARY OUTCOMES:
MK0217 will be safely tolerated

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Hooper M, Faustino A, Reid IR, Hosking D, Gilchrist NL, Selby P, Wu M, Salzmann G, West J, Leung A. Randomized, active-controlled study of once-weekly alendronate 280 mg high dose oral buffered solution for treatment of Paget's disease. Osteoporos Int. 2009 Jan;20(1):141-50. doi: 10.1007/s00198-008-0639-6. Epub 2008 Jun 7. PMID 18536953